CLINICAL TRIAL: NCT04059497
Title: Efficacy of a Short-bout Handgrip Exercise Intervention for Reducing Nicotine Craving in Tobacco Users: a Pilot Randomized Controlled Trial
Brief Title: Short-bout Handgrip Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Handgrip pilot
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking (Tobacco) Addiction
Keywords: Craving; Smoking urge; Withdrawal; Nicotine; Exercise; Isometric; Handgrip
MeSH Terms: conditions — Smoking; Behavior, Addictive; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The exercise group will receive a 10-minute exercise intervention.
  Interventions: Behavioral: Exercise condition
- Healthy diet group (Experimental): The healthy diet group (control) will receive a 10-minute healthy-diet intervention.
  Interventions: Behavioral: Healthy diet condition

INTERVENTIONS:
Behavioral: Exercise condition — Each participant in the intervention group can freely choose a handgrip of strength from 10 to 25kg which can be gripped with adequate grip strength. The PI will play the short video (5 minutes, www.youtube.com/watch?v=mZex2Wwy3fU) about the 10s-E for the participant, including (1) rapid grip-and-release the handgrip for at least 30 times in 10seconds in each hand, and (2) short-bout hand pushing and pulling exercises without handgrip. During the video, participants are asked to follow the 10s-E demonstrated by the medical professor. After the video, the PI will guide the participant to repeat the 10s-E for 5 times within the next 5 minutes. If participants feel pain in their hands, they can slow down the exercise. Between each exercise set, rest time for 10-20 seconds will be allowed. After practicing all these exercises, participants are asked to complete a post-intervention questionnaire
  Arms: Exercise group
Behavioral: Healthy diet condition — The control group will watch two videos on healthy diet (https://www.youtube.com/watch?v=w_u4BYV2Okc). Similar to the 10s-E condition, they will complete a post-intervention questionnaire after the two videos.
  Arms: Healthy diet group

SUMMARY:
This study aims to examine the effect of practicing short-bout handgrip and isometric exercises on nicotine craving, smoking urges and withdrawal symptoms in adult smokers undergoing acute tobacco abstinence. The study is a randomized controlled trial to test the effect of practicing a set of short-bout exercises (10-second exercise) on reducing nicotine craving and withdrawals. Smokers, who have been abstinent from tobacco use for 9 hours, will join a guided exercise session using 10s-E or a healthy-diet (HD, control) intervention session, and complete a craving assessment before and 2 assessments after the respective intervention session. Primary outcomes will be nicotine craving, smoking urges and withdrawal symptoms.

DETAILED DESCRIPTION:
The study is a randomized controlled trial to test the effect of practicing a set of short-bout exercises (10-second exercise) on reducing nicotine craving and withdrawals. Smokers, who have been abstinent from tobacco use for 9 hours, will join a guided exercise session using 10s-E or a healthy-diet (HD, control) intervention session, and complete a craving assessment before and 2 assessments after the respective intervention session.

1. Target subjects

   At recruitment stage (hotspot or telephone follow-up), smokers with the following inclusion criteria (Appendix 1) will be invited to participate in an intervention and assessment session:
   * Consume 10+ traditional cigarettes a day
   * Aged 18 years or above
   * Able to communicate in Cantonese
   * Self-reported no serious injury of hands and arms
   * Self-reported no mental illnesses

   Before the intervention and assessment session, the invited participants will be assessed with the following eligibility criteria:
   * Self-reported no smoking in past 9 hours before the intervention session
   * Exhaled carbon monoxide <= 15 parts per million (ppm) or reduced by at least 50% compared to that measured at recruitment stage
2. Procedures Our recruitment staff (research assistants or student helpers) will approach smokers at the outdoor smoking hotspots, and introduce the RCT to the smokers. Potential participants will be assessed with the eligibility criteria, and asked to test their exhaled carbon monoxide with a Bedfort Smokerlyzer to confirm their smoking status. If eligible, they will be asked to participate in the intervention and assessment session of this RCT.

   Our telephone interviewers of other smoking cessation trials, which have similar eligibility criteria as the present trial, will ask their participants during their telephone interviews if they currently consume 10 cigarettes or more a day and other eligibility criteria. If eligible, they will also be invited to participate in the intervention and assessment session of this RCT.

   If all these participants agree to participate, the recruitment staff will arrange an intervention and assessment session for these participants, and request them to be abstinence from tobacco products for at least 9 hours before joining the intervention and assessment session.

   At the intervention and assessment session, the principle investigator (PI) will firstly measure the exhaled carbon monoxide and ask if the participant has been abstinent for 9 hours. If eligible, they will provide a written consent (Appendix 2), complete a baseline questionnaire (Appendix 3) (administered by the PI), and will be allocated randomly to one of two conditions: exercise or healthy-diet. All intervention and assessments will take around 40 minutes to complete. All participants will be given HK$350 shopping vouchers after completing all intervention and assessments.
3. Interventions: Exercise condition Each participant in the intervention group can freely choose a handgrip of strength from 10 to 25kg which can be gripped with adequate grip strength. The PI will play the short video (5 minutes, www.youtube.com/watch?v=mZex2Wwy3fU) about the 10s-E for the participant, including (1) rapid grip-and-release the handgrip for at least 30 times in 10seconds in each hand, and (2) short-bout hand pushing and pulling exercises without handgrip. During the video, participants are asked to follow the 10s-E demonstrated by the medical professor. After the video, the PI will guide the participant to repeat the 10s-E for 5 times within the next 5 minutes. If participants feel pain in their hands, they can slow down the exercise. Between each exercise set, rest time for 10-20 seconds will be allowed. After practicing all these exercises, participants are asked to complete a post-intervention questionnaire (Appendix 4a, administered by a RA blinded to group allocation).
4. HD intervention (Control) The control group will watch two videos on healthy diet (https://www.youtube.com/watch?v=3v1vF_zrpAc and https://www.youtube.com/watch?v=w_u4BYV2Okc). Similar to the 10s-E condition, they will complete a post-intervention questionnaire after the two videos (Appendix 4b, administered by a RA blinded to group allocation).
5. 15-minute follow-up After the post-intervention measurement, both groups are asked to watch another 10-minute of health education videos about nicotine craving (https://www.youtube.com/watch?v=NpbxHj3_qns) and healthy diet ( https://www.youtube.com/watch?v=V4wyRsl8mls), and then complete another set of post-intervention questionnaire (Appendix 5, administered by a RA blinded to group allocation).
6. Outcomes Socio-demographic characteristics, smoking history and the Fagerström Test for Nicotine Dependence (FTND) [18] will be collected at the recruitment stage. At the intervention and assessment session, nicotine craving, smoking urges and withdrawal symptoms are assessed to examine the physiological effect at baseline. Nicotine craving will be assessed with a 7-point (1-not at all, 4-somewhat, 7-extremely) scale item: "How strong is your desire to smoke right now" (West & Hajek, 2004). Smoking urge will be assessed with the 10-item Questionnaire of Smoking Urges-Brief (QSU-brief) (Yu et al., 2010). Withdrawal symptoms were measured with Mood and Physical Symptoms Scale (MPSS), including 7 components: 'irritable', 'restless', 'hungry', 'poor concentration', 'stress', 'tension', and 'depressed' (West & Hajek, 2004). Respondents can select 1 option from 5 levels (1=strongly disagree, 5=strongly agree) in each component.

   The follow-up questionnaire also includes the following questions on the satisfaction of the intervention: (1) How much would you like the intervention video? (Scale 1-5; 1 indicates strongly dislike and 5 indicates strongly like); (2) How much do you understand the intervention? (Scale 0-10; 0 indicates totally not understand it and 10 indicates totally understand it); (3) Would you agree that the intervention help quitting? (Scale 1-5; 1 indicates totally disagree and 5 indicates totally agree); (4) Are you confident to do 10s-E (exercise group) / have healthy diet (diet group)? (Scale 0-10; 0 indicates totally no confidence and 10 indicates strongly confident); (5) Do you agree you have a real plan to quit with 10s-E (exercise group) / healthy diet (diet group)? (Scale 0-10; 0 indicates strongly disagree and 10 indicates strongly agree); (6) Do you think quitting by 10s-E (exercise group) / healthy diet (diet group) is difficult? (Scale 0-10; 0 indicates totally no difficulty and 10 indicates strongly difficult); (7) Will you introduce this video to other people? Options are yes or no; (8, exercise group only) Have you followed the exercise demonstration just now in the video? Options include "Not followed totally", "I followed a little bit", "I followed most of all", and "I followed all"; and (9) Do you agree that 10s-E (exercise group) / health diet (diet group) reduced their craving (Scale 1-5; 1 indicates strongly disagree and 5 indicates strongly agree).
7. Research hypothesis The exercise group will have a significantly greater decline of the craving, smoking urges and withdrawal than the control group assessed post-intervention and 15 minutes after the intervention.
8. Effect size estimation The sample size calculation is based on the score of desire to smoke (Scale 1-7). Assuming the group difference in mean change of smoking desire is 0.75 (Ussher et al., 2009), a significance level of 1%, statistical power 90%, a sample size of 30 participants (15 each group) is needed to detect a difference between the two groups.
9. Randomization, allocation concealment and blinding Simple individual randomization method by sequentially numbered, opaque sealed envelopes (SNOSE) will be used to ensure the counselors and the participants will be blinded from the allocation sequence before the group allocation (Chan et al., 2013; Doig & Simpson, 2005). The primary investigator will prepare about 50 identical, opaque, sealed, A5-sized envelops, with a unique 3-digit number on the cover of each envelope as an identifier. Then he will create a random sequence list of the intervention or control group, and each group allocation will be sequentially numbered that is matched with the envelope identifier. A paper indicating the treatment condition will be inserted into each envelop, according to the random sequence list.

   Both the PI and the participants are not blinded from the behavioral intervention, but the outcome assessors (HKU research staff) at the 2 post-intervention follow-up are blinded from the group assignment.
10. Drop-out Participants can choose to drop out from the RCT during the study period, without any penalties or administrative procedures. If the participants refuse to continue the intervention during the intervention and assessment session, the reasons of the drop-out will be documented by the counselor and reported to the HKU research staff on the same day. The envelopes of the drop-out participants will not be re-used for other participants.
11. Statistical analysis Data will be entered into SPSS for Windows (version 20) for analysis. By intention-to-treat (ITT) analysis and worst case scenario, participants who lost to follow-up or refused the follow-up will be treated as smokers. Descriptive statistics including frequency, percentage, and mean will be used to summarize the outcomes and other variables. For the desire to smoke, QSU-brief and MPSS, linear mixed models which allow for multiple observations between subjects and account for clustering of data within subjects will be used. Both the main effect (group allocation) and interaction effect (group X time) will be analyzed.

ELIGIBILITY:
At recruitment stage (hotspot or telephone follow-up), smokers with the following inclusion criteria (Appendix 1) will be invited to participate in an intervention and assessment session:

* Consume 10+ traditional cigarettes a day
* Aged 18 years or above
* Able to communicate in Cantonese
* Self-reported no serious injury of hands and arms
* Self-reported no mental illnesses

Before the intervention and assessment session, the invited participants will be assessed with the following eligibility criteria:

* Self-reported no smoking in past 9 hours before the intervention session
* Exhaled carbon monoxide <= 15 parts per million (ppm) or reduced by at least 50% compared to that measured at recruitment stage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Nicotine craving | Baseline, immediate after intervention, 15-minute follow-up
  How strong is your desire to smoke right now (Scale 1-7)
Smoking urge | Baseline, immediate after intervention, 15-minute follow-up
  10-item Questionnaire of Smoking Urges-Brief
Withdrawal sysmptoms | Baseline, immediate after intervention, 15-minute follow-up
  Mood and Physical Symptoms Scale

CONTACTS AND LOCATIONS:
Overall Officials: Derek Cheung, PhD, Principal Investigator — School of Nursing, HKU
Locations (1):
- Tung Wah Group of Hospitals, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data are available upon request made to the principal investigator.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Zhang MJ, Cheung YTD, Wang Q, Cheng CCW, Luk TT, He WJ, Wang MP, Lam TH. Efficacy of simple and very brief handgrip and isometric exercises for reducing withdrawal symptoms in cigarette smokers: A pilot randomized controlled trial. Tob Induc Dis. 2024 May 24;22. doi: 10.18332/tid/187839. eCollection 2024. PMID 38800350